CLINICAL TRIAL: NCT01173731
Title: An Open-label Treatment Study to Evaluate the Safety, Tolerability and Efficacy of AFQ056 in Parkinson's Patients With L-dopa Induced Dyskinesias
Brief Title: Open Label, Safety, Tolerability and Efficacy of AFQ056 in Parkinson's Patients With L-dopa Induced Dyskinesias
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CAFQ056A2217; 2010-019418-25 (EudraCT Number)
Record Dates: First submitted 2010-07-28; First posted 2010-08-02 (Estimated); Last update posted 2020-12-23 (Actual); Status verified 2017-03

CONDITIONS: Parkinson Disease; Dyskinesia, Drug-Induced; Levodopa
Keywords: Parkinson Disease; L-dopa; Levodopa; Dyskinesia; involuntary movement; motor complication
MeSH Terms: conditions — Parkinson Disease; Dyskinesia, Drug-Induced; Dyskinesias | interventions — mavoglurant

ARMS (1):
- AFQ056 (Experimental)
  Interventions: Drug: AFQ056

INTERVENTIONS:
Drug: AFQ056

SUMMARY:
The purpose of this study is to generate long-term safety, tolerability and efficacy data for AFQ056 in patients who have participated in and completed any AFQ056 phase II study in PD-LID (Parkinson's disease, L-dopa induced dyskinesias).

ELIGIBILITY:
Inclusion Criteria:

* Outpatients with Parkinson's disease (PD), treated with L-Dopa, experiencing dyskinesias who have been eligible for, participated in and completed an AFQ056 phase II core study.

Exclusion Criteria:

* Surgical treatment for PD
* Cancer within the past 5 years (other than localized skin cancer and prostate cancer that has been effectively treated)
* Advanced, severe or unstable disease (other than PD) that may interfere with the study outcome evaluations

Other protocol-defined inclusion/exclusion criteria may apply

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2010-10; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Incidence and severity of AEs/SAEs, changes in vital signs, lab assessments and ECGs, in cognitive function (MMSE), psychiatric symptoms (SCOPA-PC), and underlying symptoms of PD (UPDRS part III, CGIC, PGIC). | 3.5 years

SECONDARY OUTCOMES:
Assessment of dyskinetic symptoms by change from baseline in mAIMS total score | 3.5 years
Investigator and patient assessment of clinical changes in dyskinetic symptoms and disability due to dyskinesia compared to baseline, as measured by the corresponding CGIC and PGIC items respectively | 3.5 years

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (22):
- United States (3):
  - Novartis Investigative Site, Sunnyvale, California
  - Novartis Investigative Site, Englewood, Colorado
  - Novartis Investigative Site, Indianapolis, Indiana
- Australia (3):
  - Novartis Investigative Site, Heidelberg, Victoria
  - Novartis Investigative Site, Parkville, Victoria
  - Novartis Investigative Site, Prahran, Victoria
- Canada (3):
  - Novartis Investigative Site, Ottawa, Ontario
  - Novartis Investigative Site, Gatineau, Quebec
  - Novartis Investigative Site, Greenfield Park, Quebec
- France (3):
  - Novartis Investigative Site, Clermont-Ferrand
  - Novartis Investigative Site, Lille
  - Novartis Investigative Site, Pessac
- Germany (7):
  - Novartis Investigative Site, Bochum
  - Novartis Investigative Site, Dresden
  - Novartis Investigative Site, Kassel
  - Novartis Investigative Site, Marburg
  - Novartis Investigative Site, München
  - Novartis Investigative Site, Stadtroda
  - Novartis Investigative Site, Tübingen
- Italy (3):
  - Novartis Investigative Site, Lido di Camaiore, LU
  - Novartis Investigative Site, Roma, RM
  - Novartis Investigative Site, Napoli

REFERENCES:
- See also: Results for CAFQ056A2217 from the Novartis Clinical Trials Website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=12724